CLINICAL TRIAL: NCT04274673
Title: The Correlation Between the Cotinine Levels in Urine and Postoperative Acute and Chronic Pain in Open Abdominal Hysterectomy Patients
Brief Title: The Correlation Between Cotinine and Postoperative Acute and Chronic Pain After Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Assoc.Prof.MD, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2017/181
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain, Acute Pain, Cotinine, Hysterectomy
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low (less 10ng/dl) (Other): Patients who have low cotinine levels (less 10ng/dl)
  Interventions: Device: measuring cotinine level
- medium (10-500ng/dl) (Other): Patients who have medium cotinine levels (less 10-500ng/dl)
  Interventions: Device: measuring cotinine level
- high (more 500ng/dl) (Other): Patients who have high cotinine levels (less 10-500ng/dl)
  Interventions: Device: measuring cotinine level

INTERVENTIONS:
Device: measuring cotinine level — Measuring of the cotinine levels

SUMMARY:
It is known that there is an association between smoking and acute/chronic pain. But it is so difficult to assess this relation with asking questions to the patients in the preoperative period. Because of that we want to measure the levels of the cotinine in the urine and later assess the correlation with acute and chronic pain in hysterectomy patients.

DETAILED DESCRIPTION:
It is well-known that smoking is very common in the public. The chronic pain after hysterectomy is 20-40%. The open abdominal hysterectomy ratio is 75% of all hysterectomy operations in our country. We know that the reasons of postoperative acute and chronic pain is multifactorial. One of them is smoking which affects the postoperative pain. The best way of measuring the level of cotinine is assesing the urine of the patient. We collect the first urine after induction.

In this study, we aimed to investigate the correlation between the levels of urine cotinine and the acute and chronic postoperative pain in hysterectomy patents.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Open abdominal hysterectomy patients

Exclusion Criteria:

* Chronic pain
* Chronic pain killer users
* Axis I psychiatric disease
* Liver disease
* Renal disease
* Drug allergy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 158 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-13 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Chronic pain: VAS score | Postoperative 3 months
  3rd month pain after hysterectomy (VAS score)

SECONDARY OUTCOMES:
Acute pain: VAS score | Postoperative 48 hours
  Postoperative 24 hrs after hysterectomy (VAS score)

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Kemal University Medicine Faculty Anesthesiology Department, Hatay, Turkey (Türkiye)

REFERENCES:
- [Background] Montbriand JJ, Weinrib AZ, Azam MA, Ladak SSJ, Shah BR, Jiang J, McRae K, Tamir D, Lyn S, Katznelson R, Clarke HA, Katz J. Smoking, Pain Intensity, and Opioid Consumption 1-3 Months After Major Surgery: A Retrospective Study in a Hospital-Based Transitional Pain Service. Nicotine Tob Res. 2018 Aug 14;20(9):1144-1151. doi: 10.1093/ntr/ntx094. PMID 28472423